CLINICAL TRIAL: NCT05338359
Title: Metrology to Enable Rapid and Accurate Clinical Measurements in Acute Management of Sepsis
Acronym: SEPTIMET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoire National de Métrologie et d'essais (Unknown); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP191016; 2021-A01612-39 (Other: ANSM)
Record Dates: First submitted 2022-01-28; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-01

CONDITIONS: Sepsis Syndrome
Keywords: Procalcitonin; Biomarkers
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sample — Blood sample of 34 mL
Other: Phone-call — Phone-call to the participant 15 days after recruitment to fix the final diagnosis

SUMMARY:
Sepsis is a life-threatening condition that arises when a dysregulated response to infection results in multi-organ dysfunction or failure. This can affect any organ, resulting in a diverse clinical presentation. Sepsis affects more than 3.4 million Europeans a year with 700,000 deaths from the condition and an additional one third of survivors dying through complications in the year following a sepsis event.

To date, biomarkers that are used to predict bacterial infection (such as CRP or lactate) are used in combination and with other clinical symptoms due to the fact that they are non-specific for sepsis. The use of such biomarkers frequently varies between hospitals or even physicians. Biomarkers such as procalcitonin (PCT) have been reported as useful for differentiating between infectious and non-infectious causes of systemic inflammatory response syndrome. Yet calibration of PCT assays is problematic due to the absence of higher order method or international standard. External quality assessment (EQA) programs have highlighted poor comparability.

This protocol is part of the international SEPTIMET project. The Emergency Department (ED) of the Pitié-Salpêtrière hospital takes part of the project with specific objectives in order to establish a large cohort of patients at very early stage sepsis (defined by Systemic Inflammatory Response Syndrome -SIRS - due to bacterial infection or the first symptoms of sepsis before septic shock, patients consulting in the first hours of the history of the disease at the emergency department) with the idea of spotting the condition before it manifests as a more serious presentation. This will measure the clinical criteria and putative biomarkers as patients progress to more serious presentation. Moreover, an expected biobank of >200 samples will be generated to provide material for the Laboratoire National de Métrologie et d'essais (LNE) in charge of analytical studies.

DETAILED DESCRIPTION:
Sepsis accounts for ~50% of intensive care bed days and can have mortality of >30%. As time to diagnosis is the critical factor in managing sepsis the recommendation for research to shorten and improve diagnosis is particularly pertinent: the window for initiating appropriate treatment is 6 hours or less. Survival is linearly correlated with time to appropriate antibiotic treatment: each hour delay increases the chance of mortality by ~7.6% making fast/accurate diagnosis essential. This fact is met by a woefully inadequate situation where today's clinicians simply do not have diagnostic tests with sufficient accuracy and speed to meet this need. This forces them to essentially guess the best antibiotic to use, which results in inadequate treatment as well as promoting antimicrobial resistance. For today's sepsis patients the reality is that they have a treatable condition that is missed due to delayed diagnosis, quickly leading to multiple organ failure and death. Delayed treatment can also affect patients who survive sepsis due to debilitating long-term effects post-sepsis including amputations, organ dysfunction (e.g. renal failure), psychological and cognitive impairment, chronic pain, tiredness and a reduced quality of life.

Procalcitonin is widely reported as a useful biochemical marker to differentiate sepsis from other non-infectious causes of systemic inflammatory response syndrome. PCT is the pro-hormone of calcitonin that is synthetized by thyroid cells. In healthy individuals, serum PCT concentrations range below 0.1 μg/L. During sepsis, many tissues and immune cells become able to secrete PCT in the serum, due to an unsolved and complex network with cytokines. Some experimental data suggests that PCT may be an actor and not only a marker of sepsis.

Serum procalcitonin (PCT) dosage is more specific for the diagnosis of bacterial infection than C-Reactive Protein (CRP). PCT levels do not increase or only slightly in non-bacterial inflammatory syndromes. PCT also provides prognostic information and risk stratification assessment in the emergency unit. Contrary to CRP, PCT levels remain low or only slightly elevated in case of inflammatory processes except in case of bacterial infection, notably during systemic disease flares and viral infection. It is currently the first-line biomarker of infection in the emergency unit.

PCT is recognised as a biomarker of bacterial infection given that PCT is upregulated after a bacterial insult. Moreover, PCT levels decrease rapidly after the end of the insult. Thus, rapid and reliable measurement of PCT is promising for the early and accurate identification of sepsis. Particularly, improving accuracy of measurements for low concentrated samples will strengthen the role of PCT as an early diagnosis biomarker. The development of a mass spectrometry based method for the quantification of PCT by improving the quantification method developed in the earlier EMPIR project 15HLT07 AntiMicroResist will support the improvement of the traceability and accuracy of measurements performed currently in clinics for the quantification of this biomarker.

Combining multiple biomarker measurements would potentially bring a strong added-value for the diagnosis of sepsis as patterns of different analytes may continue to specify sepsis should any one biomarker fail. Thus, the multiplex method that will be developed will ameliorate the diagnostic accuracy by simultaneously monitoring a panel of sepsis biomarkers. This might pave the way towards the development of new rapid diagnosis assays targeting several protein biomarkers by in vitro diagnostics (IVD) providers.

The work performed in previous EMPIR project 15HLT07 showed the technical difficulties (sample preparation, limit of detection, robustness of the measurement) to obtain an internationally agreed reference system for the low concentrations of PCT in matrix samples. Within the new SEPTIMET project, an International System of Unit (SI) traceable higher order reference method will be developed allowing measurement over the entire range of PCT concentration. Additionally quality control materials being developed will allow improvements in the evaluation of accuracy and comparability of results across different analytical platforms to define robust clinical decision limits. Establishing this new reference system will enable PCT measurements in clinics to be accurate and reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Patient attending the ED, suspected to have bacterial infection by the emergency physician after clinical exam, and requiring a blood sampling in the ED,
* Ages Eligible for Study: 18 to 100 years-old
* PCT prescribed by physician
* Non-opposition obtained from the patient or, if not capable to express his/her non-opposition, a trustworthy person, a family member or a close relative.
* For the collection of biological samples and subsequent genetic analysis, informed consent signed by the patient

Exclusion Criteria:

* Patient minor under 18
* Pregnancy
* Anticipated difficulties for the follow-up at D15 (homeless...)
* Previously enrolled in this study (i.e. subjects may not be enrolled more than
* Patient with positive serology (HIV, HBV, HCV…)
* Patient without Social Security
* Refusal to participate from the patient or, if not capable to express himself/herself, a trustworthy person, a family member or a close relative
* Patient under guardianship or curatorship
* Patient deprived of their liberty by a judicial or administrative decision

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the ED, suspected to have bacterial infection by the emergency physician after clinical exam, and requiring a blood sampling.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Procalcitonin (PCT) measurements in serum assessed by Isotope dilution coupled to high-performance liquid chromatography and mass spectrometry | Day 0

SECONDARY OUTCOMES:
Procalcitonin (PCT) measurements in serum assessed by standard immunoassay technique | Day 0
Calculation of Systemic Inflammatory Response Syndrome (SIRS) score | Day 0
  This score is based of the assessment of 4 parameters : temperature, heart rate, respiratory rate and white bood cells count. The score is rated from 0 to 4, with 4 being the worst score.
Calculation of quick Sequential Organ Failure Assessment (qSOFA) score | Day 0
  This score is based of the assessment of 3 parameters : mentation, systolic blood pressure and respiratory rate. The score is rated from 0 to 3, with 3 being the worst score.
Calculation of Sequential Organ Failure Assessment (SOFA) score | Day 0
  This score is based of the assessment of 6 organ systems: respiratory system, coagulation system, liver system, cardiovascular system, central nervous system, renal system. Each system is rated from 0 to 4 (specific definiton for each system evaluation are provided), with 4 being the worst score. The final SOFA score corresponds to the sum of the 6 systems.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia VELLY, MD, Principal Investigator — GH Pitié Salpêtrière - Charles Foix
Locations (1):
- Pitié-Salpêtrière hospital / Emergency Department, Paris, France